CLINICAL TRIAL: NCT05778253
Title: Circulating Tumor DNA (ctDNA) Dynamic Monitoring Plus Artificial Intelligence (AI)-Based Pathology Predict the Efficacy of Chemoimmunotherapy in Resectable Lung Squamous Cell Carcinoma (LSCC)
Brief Title: The Role of ctDNA Testing Plus AI-based Pathology in Resectable LSCC
Status: Recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Shanghai OrigiMed Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Liu Wenliang, Professor, Second Xiangya Hospital of Central South University
Other Study IDs: LYF2022198
Record Dates: First submitted 2023-02-23; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Lung Squamous Cell Carcinoma
MeSH Terms: interventions — Exome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pretreatment biopsy tissue for WES testing Peripheral blood tissue for ctDNA testing
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with lung Squamous Cell Carcinoma receiving neoadjuvant chemoimmunotherapy
  Interventions: Diagnostic Test: WES and ctDNA detection

INTERVENTIONS:
Diagnostic Test: WES and ctDNA detection — WES and ctDNA detection

SUMMARY:
The goal of this observational study is to explore whether ctDNA dynamic monitoring plus AI-based pathology can more effectively predict the therapeutic effect of neoadjuvant chemoimmunotherapy for resectable lung squamous cell carcinoma, so as to accurately guide clinical diagnosis and treatment.

DETAILED DESCRIPTION:
This study is a single-center, observational, non-interventional, prospective study. 50 patients diagnosed with lung squamous cell carcinoma receiving neoadjuvant chemoimmunotherapy (ranging 2 to 4 cycles) will be planned to be enrolled in the study. Pre-treatment biopsy tissues of enrolled patients will be collected for whole exon sequencing (WES) testing, and personalized detection panel will be customized based on WES testing results. Peripheral blood will be collected 1 day before each cycle of neoadjuvant therapy, 1 day before surgery, 3 days after surgery, and 3 weeks after surgery for ctDNA testing. In addition, the prediction model of AI-based pathology will be constructed by AI deep learning based on pathological sections of pre-treatment biopsy tissues. All inclued patients will be regularly followed up for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology or cytology confirmed the lung squamous cell carcinoma
* Age ranging from 18 to 75
* Agree to participate in this study and sign an informed consent form
* Treatment-naive tumor
* According to the American Joint Committee on Cancer (AJCC) eighth edition of the Lung Cancer Staging Manual, the clinical stage is stage II-IIIb resectable or potentially resectable tumor
* Sufficient tissue/blood samples are available to meet research requirements
* The ECOG PS score is 0-1

Exclusion Criteria:

* Patients who cannot understand the content of the experiment and cannot cooperate, and those who refuse to sign the informed consent form
* Non-squamous NSCLC
* Unresectable IIIa-IIIb tumor
* Patients with solid organ or blood system transplantation
* Previous use of CTLA-4, PD-1, or PD-L1 immune checkpoint inhibitors
* Patients with interstitial lung disease
* Patients with acute or chronic infectious disease
* Pregnant and lactating women
* Patients who have undergone other clinical drug trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Resectable or potentially resectable stage II-IIIb lung squamous cell carcinoma patients receiving neoadjuvant chemoimmunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-23 (Estimated); Primary Completion 2028-09-23 (Estimated); Study Completion 2029-09-23 (Estimated)

PRIMARY OUTCOMES:
Pathologic completet response (pCR) rate | Up to 1 year
  pCR rate is defined as the percentage of participants having an absence of residual tumor cells in resected lung specimens and lymph nodes following completion of neoadjuvant therapy.
ctDNA resolution | Up to 2 years
  ctDNA resolution is defined as the change or resolution in tumor-derived DNA found in the bloodstream from diagnosis to after neoadjuvant therapy and after surgery, correlated with pathologic complete response (pCR)
Development of computer algorithm to identify pCR features | From retrospective data collection to algorithm development (6 month)
  Development of computer algorithm to identify pCR features
Validation of computer algorithm to identify pCR features | From prospective data collection to algorithm validation (6 months)
  Validation of computer algorithm to identify pCR features

SECONDARY OUTCOMES:
Major pathological response (MPR) rate | Up to 1 year
  MPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and resected lymph nodes following completion of neoadjuvant therapy.
Objective response rate(ORR) | Up to 1 year
  The proportion of patients achieved complete or patial remission(Imageological) according to RECIST 1.1 prior to definitive surgery.
Adverse events (AEs) | Up to 5 years
  Number of participants experiencing AEs will be recorded. An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Perioperative complications rate | Up to 3 years
  Number of participants experiencing perioperative complications will be recorded.
Health-related Quality of Life | Up to 5 years
  Health-related Quality of Life will be assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) version 3.0, the EORTC Quality of Life Questionnaire in Lung Cancer (EORTC QLQ-LC13), and the European Quality of Life 5 Dimensions (EQ-5D) questionnaire.
Perioperative pain evaluation | Up to 3 years
  Perioperative pain evaluation assessed by a numeric rating scale (NRS)
Disease free survival (DFS) | Up to 5 years
  From the date of surgery to any of the following events: disease progression, disease recurrence or death from any cause.
Overall survival (OS) | Up to 5 years
  From the date of participated in study to the date of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Thoracic Surgery, Second Xiangya Hospital of Central South University, China, Changsha, Hunan, China